CLINICAL TRIAL: NCT06335771
Title: Harnessing Macrophage Lysosomal Lipid Metabolism in Obesity-Associated Diseases
Brief Title: Harnessing Macrophage Lysosomal Lipid Metabolism in Obesity
Acronym: ATM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bettina Mittendorfer (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Washington University School of Medicine (Other)
Responsible Party: Sponsor-Investigator, Bettina Mittendorfer, Senior Associate Dean for Research; Professor, Medicine & Nutrition; NextGen Director of Clinical and Translational Sciences Unit, University of Missouri-Columbia
Organization: University of Missouri-Columbia (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2098077; R01DK131188 (NIH)
Record Dates: First submitted 2024-03-14; First posted 2024-03-28 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Obesity; Nonalcoholic Fatty Liver; Diabetes Type 2; Healthy
MeSH Terms: conditions — Obesity; Non-alcoholic Fatty Liver Disease; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Lean Individuals (No Intervention): No intervention will be administered.
- Metabolically abnormal obese Individuals (obesity with normoglycemia and abnormal liver fat content) (Experimental): Participants will undergo a dietary weight loss intervention to achieve 10% weight loss over about 6 months.
  Interventions: Other: Dietary consultation weight loss intervention
- Metabolically normal obese Individuals (obesity with normoglycemia and normal liver fat content) (Experimental): Participants will undergo a dietary weight loss intervention to achieve 10% weight loss over about 6 months.
  Interventions: Other: Dietary consultation weight loss intervention
- Individuals with Type 2 Diabetes Mellitus (Experimental): Participants will undergo a dietary weight loss intervention to achieve 10% weight loss over about 6 months.
  Interventions: Other: Dietary consultation weight loss intervention

INTERVENTIONS:
Other: Dietary consultation weight loss intervention — Participants will meet with a member of the study team biweekly for about 6 months.
  Arms: Individuals with Type 2 Diabetes Mellitus; Metabolically abnormal obese Individuals (obesity with normoglycemia and abnormal liver fat content); Metabolically normal obese Individuals (obesity with normoglycemia and normal liver fat content)

SUMMARY:
The goal of this study is to evaluate the role of transcription factor EB (TFEB) in adipose (fat) tissue macrophages (ATM) in regulating adipose tissue and systemic metabolic function in obesity. The investigators will assess the differences in ATM lipid metabolism in people with metabolically abnormal obesity and lean individuals.

Both groups will have:

* screening visit
* imaging (body composition testing - dual-energy x-ray absorptiometry (DEXA) scans, magnetic resonance imaging [MRI] and magnetic resonance spectroscopy [MRS] scans)
* Overnight visit with intravenous infusion (IV), muscle, and fat tissue biopsies Participants with obesity will complete meetings with study team members for a weight loss intervention to achieve a 10% body weight loss.

ELIGIBILITY:
Inclusion Criteria :

* age: ≥18 but ≤70 years
* not pregnant or breastfeeding
* weight stable and sedentary before enrollment
* no use tobacco products, excessive amounts of alcohol, or dietary supplements, or medications known to or suspected to affect glucose and lipid metabolism (aside from certain medications used to treat diabetes in the metabolically abnormal obesity [MAO]-Type 2 Diabetes group)
* no evidence of significant organ system dysfunction or disease (e.g. chronic severe kidney disease, cancer)
* participants must fulfil all of the following group-specific inclusion criteria below:

Lean group:

* Body mass index (BMI) ≥18.5 but <25.0 kg/m2
* Intrahepatic triglyceride (IHTG) content <5%
* fasting blood glucose concentration: <100 mg/dl
* blood glucose concentration 2 h after a 75 g oral glucose challenge: <140 mg/dl
* Hemoglobin A1C (HbA1c) <5.7 %

Metabolically normal obesity (MNO) group:

* BMI ≥30.0 but <45.0 kg/m2
* IHTG content <5%
* fasting blood glucose concentration: <100 mg/dl
* blood glucose concentration 2 h after a 75 g oral glucose challenge: <140 mg/dl
* HbA1c <5.7 %

Metabolically abnormal obesity (MAO)-insulin resistance and non-alcoholic fatty liver disease (NAFLD) group:

* BMI ≥30.0 but <45.0 kg/m2
* IHTG content >7.5%
* fasting blood glucose concentration: ≥100 but <126 mg/dl
* blood glucose concentration 2 h after a 75 g oral glucose challenge: ≥140 but <200 mg/dl
* HbA1c: ≥5.7 but <6.4 %

MAO-type 2 diabetes group:

* BMI ≥30.0 but <45.0 kg/m2
* clinical diagnosis of type 2 diabetes or fasting blood glucose concentration >126 mg/dl or blood glucose concentration 2 h after a 75 g oral glucose challenge>200 mg/dl or HbA1c >6.4 % without medication if not diagnosed and medically treated for diabetes

Exclusion Criteria:

- Individuals that do not meet all inclusion Criterion

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2028-03 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Insulin sensitivity assessed as insulin-mediated glucose disposal during a hyperinsulinemic-euglycemic clamp procedure. | up to 6 months after the intervention
24-hour plasma glucose concentration | up to 6 months after the intervention
Macrophage isolation in adipose tissue biopsy | up to 6 months after the intervention
  macrophage gene expression using RNA sequencing and fluorescent activated cell sorting (FACS)
Macrophage isolation in skeletal muscle tissue | up to 6 months after the intervention
  macrophage gene expression using RNA sequencing and fluorescent activated cell sorting (FACS)

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Mittendorfer, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri School of Medicine, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No